CLINICAL TRIAL: NCT04736212
Title: Assessment of Breathing Using an Under-bed Weighing Scale
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Chiba University (Other)
Responsible Party: Principal Investigator, Maximilian S Schaefer, Assistant Professor of Anesthesia, Beth Israel Deaconess Medical Center
Other Study IDs: 2020P001209
Record Dates: First submitted 2021-01-29; First posted 2021-02-03 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Respiratory Complication; Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bed sensor monitoring system — Respiratory patterns in the post-anesthesia care unit will be assessed using a validated, modified under bed weighing scale placed under the patient's bed in the PACU.

SUMMARY:
The aim of this study is to assess the capability of a modified under bed weighing scale (contact-free unconstrained respiratory monitor, BSS) to predict postoperative pulmonary complications in high-risk surgical patients.

The study is designed to test the hypothesis that abnormal breathing measured by a modified under bed weighing scale predicts postoperative pulmonary complications within 7 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Undergoing non-cardiac surgery under general anesthesia.
3. Score ≥ 25 in the risk prediction score (Table1)

Exclusion Criteria:

1. Ambulatory (outpatient) surgery
2. Transfer directly to the ICU
3. Remain intubated/ planned to remain intubated after surgery
4. Pregnant patients: as detected by patient self-reporting of diagnosed by preoperative pregnancy testing according to institutional policies at BIDMC.
5. Patients enrolled in other interventional studies which could confound the primary endpoint.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We anticipate that our study population will reflect the normal distribution of race and gender of patients presenting for surgeries at BIDMC.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Postoperative pulmonary complications | First 7 postoperative days
  atelectasis, pneumonia, acute respiratory distress syndrome, pulmonary aspiration, re-intubation, unprecedented non-invasive ventilation, unplanned ICU admission, or re-admission to the hospital due to respiratory complication.

SECONDARY OUTCOMES:
Postoperative pulmonary complications | First 3 postoperative days
  atelectasis, pneumonia, acute respiratory distress syndrome, pulmonary aspiration, re-intubation, unprecedented non-invasive ventilation, unplanned ICU admission, or re-admission to the hospital due to respiratory complication.
Major adverse Cardiovascular events | First 7 postoperative days
  death, myocardial infarction, coronary revascularization, stroke, and heart failure.
Hospital length of stay | 30 days after surgery
  Duration from surgery to hospital discharge
Adverse discharge disposition | 30 days after surgery
  lost of ability to live independently: adverse discharge disposition to a skilled nursing facility or in-hospital mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Result] de la Gala F, Pineiro P, Reyes A, Vara E, Olmedilla L, Cruz P, Garutti I. Postoperative pulmonary complications, pulmonary and systemic inflammatory responses after lung resection surgery with prolonged one-lung ventilation. Randomized controlled trial comparing intravenous and inhalational anaesthesia. Br J Anaesth. 2017 Oct 1;119(4):655-663. doi: 10.1093/bja/aex230. PMID 29121283
- [Result] Andersen LW, Berg KM, Chase M, Cocchi MN, Massaro J, Donnino MW; American Heart Association's Get With The Guidelines((R))-Resuscitation Investigators. Acute respiratory compromise on inpatient wards in the United States: Incidence, outcomes, and factors associated with in-hospital mortality. Resuscitation. 2016 Aug;105:123-9. doi: 10.1016/j.resuscitation.2016.05.014. Epub 2016 May 30. PMID 27255952
- [Result] Khanna AK, Overdyk FJ, Greening C, Di Stefano P, Buhre WF. Respiratory depression in low acuity hospital settings-Seeking answers from the PRODIGY trial. J Crit Care. 2018 Oct;47:80-87. doi: 10.1016/j.jcrc.2018.06.014. Epub 2018 Jun 18. PMID 29936327
- [Result] Boden I, Skinner EH, Browning L, Reeve J, Anderson L, Hill C, Robertson IK, Story D, Denehy L. Preoperative physiotherapy for the prevention of respiratory complications after upper abdominal surgery: pragmatic, double blinded, multicentre randomised controlled trial. BMJ. 2018 Jan 24;360:j5916. doi: 10.1136/bmj.j5916. PMID 29367198
- [Result] Isono S, Nozaki-Taguchi N, Hasegawa M, Kato S, Todoroki S, Masuda S, Iida N, Nishimura T, Noto M, Sato Y. Contact-free unconstraint respiratory measurements with load cells under the bed in awake healthy volunteers: breath-by-breath comparison with pneumotachography. J Appl Physiol (1985). 2019 May 1;126(5):1432-1441. doi: 10.1152/japplphysiol.00730.2018. Epub 2019 Feb 14. PMID 30763161
- [Result] Schaefer MS, Eikermann M. Contact-free respiratory monitoring using bed wheel sensors: a valid respiratory monitoring technique with significant potential impact on public health. J Appl Physiol (1985). 2019 May 1;126(5):1430-1431. doi: 10.1152/japplphysiol.00198.2019. Epub 2019 Mar 28. No abstract available. PMID 30920886
- [Result] Abbott TEF, Fowler AJ, Pelosi P, Gama de Abreu M, Moller AM, Canet J, Creagh-Brown B, Mythen M, Gin T, Lalu MM, Futier E, Grocott MP, Schultz MJ, Pearse RM; StEP-COMPAC Group. A systematic review and consensus definitions for standardised end-points in perioperative medicine: pulmonary complications. Br J Anaesth. 2018 May;120(5):1066-1079. doi: 10.1016/j.bja.2018.02.007. Epub 2018 Mar 27. PMID 29661384
- [Result] Choi BG, Rha SW, Yoon SG, Choi CU, Lee MW, Kim SW. Association of Major Adverse Cardiac Events up to 5 Years in Patients With Chest Pain Without Significant Coronary Artery Disease in the Korean Population. J Am Heart Assoc. 2019 Jun 18;8(12):e010541. doi: 10.1161/JAHA.118.010541. Epub 2019 Jun 12. PMID 31185781